CLINICAL TRIAL: NCT06939985
Title: Cardiometabolic Risk Factors and Clinical Outcomes in Heart Failure: An Observational Cohort Study
Brief Title: Cardiometabolic evalUation REgistry of Heart Failure
Acronym: CURE-HF
Status: Recruiting | Type: Observational
Sponsor: Ruijin Hospital (Other)
Responsible Party: Principal Investigator, RUIYAN ZHANG, M.D., Ph.D., FACC, FESC, Ruijin Hospital
Other Study IDs: RJH-CUREHF
Record Dates: First submitted 2025-04-08; First posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Heart Failure; Metabolic Cardiovascular Syndrome; Metabolic Diseases
Keywords: heart failure; cardiometabolic risk factors; epicardial adipose tissue; cardiac remodeling; heart failure phenotypes; major adverse cardiovascular events
MeSH Terms: conditions — Heart Failure; Metabolic Syndrome; Metabolic Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a combined retrospective-prospective observational cohort study investigating the role of systemic and local cardiometabolic risk factors in cardiac structural/functional remodeling and clinical outcomes among heart failure (HF) patients. The study integrates retrospective clinical data (from the past 10 years) and prospective longitudinal follow-up (5 years) of HF patients across HF with reduced (HFrEF), mildly-reduced (HFmrEF), preserved (HFpEF) and improved ejection fraction (HFimpEF) phenotypes. Systemic metabolic factors (e.g., blood lipid profiles, glycemic levels, insulin resistance) and local factors (e.g., epicardial adipose tissue [EAT], perivascular adipose tissue [PVAT]) will be analyzed for their associations with changes in cardiac geometrics and function, dynamic transitions between HF phenotypes, as well as the occurrence of major adverse cardiovascular events (MACEs). The study seeks to advance risk stratification by integrated evaluation of cardiometabolic profiles so as to refine personalized cures in HF management.

DETAILED DESCRIPTION:
This is a combined retrospective-prospective observational cohort study aiming to elucidate the interplay between systemic/localized cardiometabolic risk factors and their impact on myocardial remodeling, cardiac function, and clinical trajectories in heart failure (HF) patients. By harmonizing retrospective clinical data spanning the past decade with a 5-year prospective longitudinal follow-up, the study encompasses all HF phenotypes, including reduced (HFrEF), mildly reduced (HFmrEF), preserved (HFpEF), and improved ejection fraction (HFimpEF), to capture the full spectrum of disease heterogeneity. Systemic metabolic dysregulation, such as dyslipidemia, impaired glucose metabolism, obesity and other metabolites assessed by mass spectrometry (MS), will be evaluated alongside localized factors, such as epicardial adipose tissue (EAT), perivascular adipose tissue (PVAT) quantified by advanced imaging modalities (cardiac MRI or CT). These factors will be correlated with changes in cardiac geometry (e.g., left ventricular mass, chamber dimensions, wall thickness) and function (e.g., ejection fraction, strain imaging, diastolic parameters), dynamic transitions between HF phenotypes (e.g., HFrEF to HFimpEF), as well as the occurrence of major adverse cardiovascular events (MACEs), defined as a composite of HF re-hospitalization and cardiovascular death. The prospective cohort will undergo standardized baseline assessments (blood biomarkers, echocardiography, cardiac CT or MRI) followed by routine clinical, biochemical and imaging evaluations at least 3-month intervals. Retrospective data will be extracted from electronic health records, including historical imaging studies, laboratory results, and event documentation, ensuring a robust sample size (target n≈3500 retrospective; n≈1200 prospective) for stratified analyses by HF phenotype, sex, and metabolic risk tertiles. Advanced statistical approaches, including multivariable regression analysis, multivariable Cox proportional hazards models and machine learning algorithms, will identify independent predictors for cardiac remodeling, functional alterations, HF phenotype transitions and MACEs. Ethical approval and informed consent are obtained for prospective participants, with retrospective data anonymized to ensure privacy. This study is expected to refine risk stratification tools by integrating metabolic imaging biomarkers and biochemical profiles, ultimately guiding personalized therapeutic cures for HF patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years
2. Chronic HF (NYHA II~IV), including:

   * HFrEF (HF with reduced ejection fraction): ① HF symptoms±signs ; ② LVEF≤40%.
   * HFimpEF (HF with improved ejection fraction): ① HF symptoms±signs; ② previous LVEF ≤ 40% and a follow-up measurement of LVEF >40%.
   * HFmrEF (HF with mildly reduced ejection fraction): ① HF symptoms±signs; ② LVEF 41%~49%.
   * HFpEF (HF with preserved ejection fraction): ① HF symptoms±signs; ② LVEF ≥50%; ③ objective evidence of cardiac structural and/or functional abnormalities consistent with the presence of LV diastolic dysfunction/raised LV filling pressures, including raised natriuretic peptide.

Exclusion Criteria:

1. Estimated survival ≤ 1 year.
2. Pregnant or lactation, or have the intention to give birth within one year.
3. Poor compliance, unable to follow-up.
4. Mental or physical status not allowing written informed consent.
5. Unwillingness to give informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is a combination of retrospective and prospective cohort. Ambulatory and hospitalized patients with chronic HF (NYHA II-IV) across all ejection fraction phenotypes are consecutively enrolled.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2015-01-01 (Actual); Primary Completion 2027-05-31 (Estimated); Study Completion 2030-05-31 (Estimated)

PRIMARY OUTCOMES:
Changes in cardiac function | 12 months
  Changes in ejection fraction (EF) measured by echocardiography or cardiac MRI at baseline and during follow-up.
Major cardiovascular events (MACEs) | 5 years
  A composite endpoint of HF re-hospitalizaion and cardiovascular death during follow-up

SECONDARY OUTCOMES:
HF re-hospitalization | 5 years
  The occurrence of protocol-adjudicated, unplanned hospitalization (≥24 hours requiring intravenous therapy for worsening HF, validated by symptomatic/hemodynamic criteria and biomarker/imaging evidence) during follow-up.
Cardiovascular death | 5 years
  The occurrence of cardiovascular death during follow-up.
All-cause mortality | 5 years
  The occurrence of death during follow-up
Dynamic transition among HF phenotypes | 12 months
  The occurrence of transition among HF phenotypes (HFrEF, HFimpEF, HFmrEF, HFpEF) measured by echocardiography or cardiac MRI at baseline and during follow-up
Changes in cardiac diastolic function | 12 months
  Changes in diastolic function (E/e' and E/A), measured by echocardiography at baseline an follow-up
Changes in cardiac regional myocardial contractile function | 12 months
  Changes in wall motion score index (WMSI) measured by echocardiography at baseline and follow-up
Changes in left ventricular strain | 12 months
  Changes in left ventricular strain measured by echocardiography or cardiac MR at baseline and during follow-up.
Changes in left atrial strain | 12 months
  Changes in left atrial strain measured by echocardiography or cardiac MR at baseline and during follow-up.
Changes in chamber dimensions | 12 months
  The changes in chamber dimensions analyzed by echocardiography or cardiac MRI at baseline and during follow-up
Changes in left ventricular mass | 12 months
  The changes in cardiac left ventricular mass analyzed by echocardiography or cardiac MRI at baseline and during follow-up.
Cardiac wall thickness | 12 months
  The changes in wall thickness analyzed by echocardiography or cardiac MRI at baseline and during follow-up.
Changes in epicardial adipose tissue (EAT) volume | 12 months
  Changes in the volume of EAT measured by cardiac CT or MRI and quantification analysis at baseline and during follow-up.
Changes in epicardial adipose tissue (EAT) density | 12 months
  Changes in the density of EAT measured by cardiac CT or MRI and quantification analysis at baseline and during follow-up.
Changes in epicardial adipose tissue (EAT) distribution | 12 months
  Changes in the distribution of EAT measured by cardiac CT or MRI and quantification analysis at baseline and during follow-up.
Changes in perivascular adipose tissue (PVAT) volume | 12 months
  Changes in the volume of PVAT measured by coronary CT angiography and quantification analysis at baseline and during follow-up.
Changes in perivascular adipose tissue (PVAT) density | 12 months
  Changes in the density of PVAT measured by coronary CT angiography and quantification analysis at baseline and during follow-up.
Changes in perivascular adipose tissue (PVAT) distribution | 12 months
  Changes in the distribution of PVAT measured by coronary CT angiography and quantification analysis at baseline and during follow-up.

CONTACTS AND LOCATIONS:
Overall Officials: Ruiyan Zhang, M.D., Ph.D., Principal Investigator — Ruijin Hospital; Xiaoqun Wang, M.D., Ph.D., Study Chair — Ruijin Hospital
Locations (1):
- Ruijin Hospital, Shanghai Jiaotong University School of Medicine, Shanghai, China